CLINICAL TRIAL: NCT04930328
Title: A Retrospective Data Collection and Analysis Study of Patients With Sickle Cell Disease (SCD) Who Have Been Treated With Oxbryta® (Voxelotor)
Brief Title: Retrospective Real World Oxbryta® Data Collection and Analysis Study
Acronym: RETRO
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: GBT440-4R1; C5341018 (Other: Alias Study Number)
Record Dates: First submitted 2021-06-04; First posted 2021-06-18 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease Registry
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Retrospective Data Collection: Retrospective Data Collection
  Interventions: Drug: Oxbryta® (voxelotor) 500-mg Tablets

INTERVENTIONS:
Drug: Oxbryta® (voxelotor) 500-mg Tablets — Patients will have received treatment with Oxbryta as prescribed by their physician at the approved dose per local prescribing information, as part of their usual care.
  Other Names: Voxelotor; Oxbryta®

SUMMARY:
The aim of this study is to collect and analyze retrospective data on Oxbryta in a real-world setting. This is a multicenter, retrospective data collection and analysis study to characterize health outcomes in approximately 300 patients with SCD who have been treated with Oxbryta as part of their usual care. Any patient with SCD who received Oxbryta treatment for at least 2 weeks as part of their usual care according to the Oxbryta US Prescribing Information (USPI) is eligible to participate. Study data from 1 year before and up to 1 year after the first dose of Oxbryta will be entered in case report forms (CRFs) via an electronic data capture (EDC) system by the study staff.

DETAILED DESCRIPTION:
The following are categories of interest in patients with SCD treated with Oxbryta:

* Clinical outcomes, as assessed by clinical and laboratory assessments of hematological parameters and end organ damage, and incidence of significant clinical events
* Healthcare resource utilization
* Health-related quality of life (HRQoL), as assessed by patient-reported outcome (PRO) measures and clinician-reported outcomes (ClinRO)

The safety objective is to assess the safety and tolerability of Oxbryta.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all the following criteria will be eligible for inclusion in this study:

1. Willing and able to provide written informed consent (ages greater or equal to 18 years) or parental/guardian consent and patient assent (age <18 years), as required by the IRB or institution or IRB, per local regulations
2. Male or female patients with documented diagnosis of SCD (all genotypes)
3. Have been treated with Oxbryta for at least 2 weeks, according to the Oxbryta USPI

Exclusion Criteria:

-

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients at each participating study site who have been treated with Oxbryta will be considered for inclusion in this study.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Change from pre-Oxbryta treatment period in Hemoglobin (Hb) | 1 year before and 1 year after the first dose of Oxbryta
Change from pre-Oxbryta treatment period in percent Reticulocytes | 1 year before and 1 year after the first dose of Oxbryta
Change from pre-Oxbryta treatment period in Absolute Reticulocytes | 1 year before and 1 year after the first dose of Oxbryta
Change from pre-Oxbryta treatment period in Bilirubin | 1 year before and 1 year after the first dose of Oxbryta
Incidence of significant SCD-related clinical events | 1 year before and 1 year after the first dose of Oxbryta
  Such as vaso-occlusive crisis (VOC), acute chest syndrome (ACS), priapism, cerebral infarcts, transient ischemic attack (TIA), leg ulcers, and measures of cardiac function and pulmonary hypertension (PH)
Change from pre-Oxbryta treatment period in incidence of unplanned clinic visits | 1 year before and 1 year after the first dose of Oxbryta
Change from pre-Oxbryta treatment period in incidence of emergency department (ED) visits | 1 year before and 1 year after the first dose of Oxbryta
Change from pre-Oxbryta treatment period in incidence of hospitalizations (including total length of stay and time in intensive care unit [ICU], if applicable) | 1 year before and 1 year after the first dose of Oxbryta
Change from pre-Oxbryta treatment period in incidence of red blood cell transfusions | 1 year before and 1 year after the first dose of Oxbryta
Incidence and severity of serious adverse events (SAEs) | 1 year before and 1 year after the first dose of Oxbryta
Incidence and severity of adverse events (AEs) of interest | 1 year before and 1 year after the first dose of Oxbryta
  Such as Rash, Diarrhea, Headache, AEs leading to Oxbryta dose modification or discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - University of Connecticut Health, Farmington, Connecticut
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Central Michigan University/Children's Hospital of Michigan, Detroit, Michigan
  - Rutgers Robert Wood Johnson Medical School Pediatric Clinical Research Center, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Parkland Health & Hospital System, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT440-4R1